CLINICAL TRIAL: NCT03938259
Title: Effect of Opioids on Ventilation in Children With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Assistant Professor of Anesthesiology, Baylor College of Medicine
Other Study IDs: H-45486
Record Dates: First submitted 2019-04-27; First posted 2019-05-06 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Depression; Obstructive Sleep Apnea
Keywords: pediatrics; opioids; obstructive sleep apnea
MeSH Terms: conditions — Respiratory Insufficiency; Sleep Apnea, Obstructive | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group; patients without obstructive sleep apnea: Children without OSA having procedures requiring endotracheal intubation and an who will receive opioids for evaluation of respiratory changes
  Interventions: Drug: Fentanyl
- Patients with known obstructive sleep apnea: Children with OSA having adenotonsillectomy for obstructive apnea will receive opioids with evaluation of respiratory changes
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — identification of respiratory parameter changes following administration of fentanyl in children with and without OSA
  Other Names: respiratory changes, CO2, RR, TV

SUMMARY:
The sole objective in this study is to evaluate if routine amounts of opioids given for tonsillectomy in children have greater amounts of respiratory depression in children with documented obstructive sleep apnea when compared with patients that do not have obstructive sleep apnea

DETAILED DESCRIPTION:
Ventilatory suppression in children following opioid administration is of obvious concern, especially following routine surgical procedures (i.e. adenotonsillectomy). It is thought that patients with obstructive sleep apnea (OSA) have increased sensitivity to opioids, and especially in opioid naïve patients. Recent evidence in adults suggests that patients with moderate to severe OSA may not predispose patients to increased opioid sensitivity in the form of respiratory depression when compared with patients that do not have OSA. It is well known that OSA in children is significantly different from OSA in adults (e.g. gender predilection, central vs. peripheral causation). The manifestation and etiologies are very different in pediatric OSA making it a vastly different disease process.

ELIGIBILITY:
Inclusion Criteria:

* tonsillectomy or adenotonsillectomy
* Ages 2 to 8 years
* Polysomnography with AHI >6 (study group)
* Polysomnography with AHI =0 or negative OSA 18 questionnaire (control group)

Exclusion Criteria:

* Ages >8 years
* Patients requiring pre-medication
* Parental refusal
* Opioid allergy/intolerance
* Patients requiring propofol for intubation
* Patients with known or suspected difficult airway
* Obesity with body mass index exceeding 30- (control group only)
* Known cardiovascular disorders
* Known pulmonary disorders aside from asthma
* Patients with chronic oxygen requirement
* History of Prematurity <35 weeks of gestation
* No recent URI
* Personal of family history of malignant hyperthermia

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We are assessing the effect of fentanyl on children with and without OSA based on the OSA 18 questionnaire and PSG resepctively. Children must be otherwise healthy as stated above in the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: adam adler, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No information about IP will be shared per the IRB

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group; Patients Without Obstructive Sleep Apnea | Patients With Known Obstructive Sleep Apnea
Started | 21 | 31
Completed | 20 | 30
Not Completed | 1 | 1
Not completed — unable to establish baseline for ventilation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group; Patients Without Obstructive Sleep Apnea | Patients With Known Obstructive Sleep Apnea | Total
Number analyzed (Participants) | 20 | 30 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.6 (1.5) | 3.6 (1.7) | 4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 14 | 19 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 13 | 20
  Not Hispanic or Latino | 13 | 17 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 14 | 23 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 30 | 50

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Depression Following Opioids
Description: Identification of respiratory depression following routine fentanyl administration by recording the respiratory rate prior to and 10 minutes following fentanyl administration
Time Frame: Mean respiratory rate % change from baseline measured 10 minutes following opioid administration
Measure: Mean (95% Confidence Interval); unit: percentage of change from baseline
Arm/Group | Control Group; Patients Without Obstructive Sleep Apnea | Patients With Known Obstructive Sleep Apnea
Number analyzed (Participants) | 20 | 30
percentage of change from baseline | -38.1 [-42.3 to -33.9] | -37.1 [-43.4 to -30.8]

2. Primary Outcome: Respiratory Depression Following Opioids
Description: Identification of respiratory depression following routine fentanyl administration by recording the tidal volume % change from baseline prior to and 10 minutes following fentanyl administration
Time Frame: mean percentage of change from baseline in tidal volume measured 10 minutes following opioid administration
Measure: Mean (95% Confidence Interval); unit: percentage of change from baseline
Arm/Group | Control Group; Patients Without Obstructive Sleep Apnea | Patients With Known Obstructive Sleep Apnea
Number analyzed (Participants) | 20 | 30
percentage of change from baseline | 6.4 [-1.2 to 13.9] | 5.4 [0.0 to 10.7]

3. Primary Outcome: Respiratory Depression Following Opioids
Description: Identification of respiratory depression following routine fentanyl administration by recording the end-tidal co2 % change from baseline prior to and 10 minutes following fentanyl administration
Time Frame: mean percentage of change from baseline in end tidal co2 measured 10 minutes following opioid administration
Measure: Mean (95% Confidence Interval); unit: percentage of change from baseline
Arm/Group | Control Group; Patients Without Obstructive Sleep Apnea | Patients With Known Obstructive Sleep Apnea
Number analyzed (Participants) | 20 | 30
percentage of change from baseline | 4.0 [1.8 to 6.1] | 2.2 [0.2 to 4.2]

ADVERSE EVENTS:
Time Frame: adverse events were collected only within the study period of ten minutes
Arm/Group | Control Group; Patients Without Obstructive Sleep Apnea | Patients With Known Obstructive Sleep Apnea
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/30
Other Adverse Events (participants affected / at risk) | 0/20 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03938259/Prot_SAP_000.pdf